CLINICAL TRIAL: NCT02573402
Title: The Effects Upon the Bladder of Transcutaneous Tibial Nerve Stimulation in Acute Traumatic Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Institute for Rehabilitation and Research (TIRR) (Unknown); Baylor College of Medicine (Other); Case Western Reserve University (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-15-0806
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injury; Neurogenic Bladder
Keywords: electric stimulation; urodynamic study
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcutaneous Tibial Nerve Stimulation (Experimental): Transcutaneous Tibial Nerve Stimulation (TTNS) applied to subjects for 2-week protocol.
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation
- Control (Sham Comparator): Sham stimulation.
  Interventions: Device: Control

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation — 10 sessions over a 2 week period of TTNS for 30 minutes. Electrodes will be placed 2 inch by 4 inch according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode, verified with rhythmic flexion of the toes secondary to stimulation of the flexor digitorum and hallicus brevis. Current intensity may vary from patient to patient and will be documented and used in the analysis.
  Arms: Transcutaneous Tibial Nerve Stimulation
Device: Control — 10 sessions over a 2 week period of TTNS sham stimulation for 30 minutes. Electrodes will be placed 2 inch by 4 inch according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode. Current intensity will be set to zero.
  Arms: Control

SUMMARY:
The purpose of this research study is to evaluate the effects upon the bladder of electric stimulation of the leg's tibial nerve in people with acute spinal cord injury with an intervention called transcutaneous tibial nerve stimulation (TTNS).

DETAILED DESCRIPTION:
In this study, TTNS will be used to help neurogenic bladder in SCI. First, acute SCI subjects which respond to TTNS will be identified as seen on urodynamic studies (USD). Then, responders will be invited to participate in a randomized control trial of a 2-week protocol of TTNS to test for safety and efficacy during inpatient rehabilitation to evaluate bladder changes based upon pre- and post- urodynamic testing, as well as 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment within 6 weeks of injury
* Neurologic level rostral to T10 (T9 and above). This is a significant neurologic level because the bladder remains innervated at these levels, without damage to the nerve cell bodies of the bladder within the spinal cord.
* Location and transportation available for follow-up appointments

Exclusion Criteria:

* History of peripheral neuropathy or premorbid symptoms of peripheral neuropathy
* Known etiologies that may cause peripheral neuropathy (i.e. diabetes mellitus, hypothyroidism, autoimmune diseases, alcoholism, hx of chemotherapy, etc.)
* History of genitourinary diagnoses (i.e. prostate hypertrophy, overactive bladder, cancer, etc.)
* Pregnancy
* History of central nervous system disorder (i.e. prior SCI, stroke, brain injury, Parkinson's disease, MS, etc.)
* Morbid obesity
* Ventilator dependent respiration
* Significant autonomic dysreflexia during baseline urodynamic study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, Principal Investigator — University of Texas at Houston Health Science Center
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Stampas A, Gustafson K, Korupolu R, Smith C, Zhu L, Li S. Bladder Neuromodulation in Acute Spinal Cord Injury via Transcutaneous Tibial Nerve Stimulation: Cystometrogram and Autonomic Nervous System Evidence From a Randomized Control Pilot Trial. Front Neurosci. 2019 Feb 19;13:119. doi: 10.3389/fnins.2019.00119. eCollection 2019. PMID 30837835

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control (Sham stimulation).
  Control: 10 sessions over a 2 week period of TTNS sham stimulation for 30 minutes. Electrodes will be placed 2 inch by 4 inch according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode. Current intensity will be set to zero.
Period: Overall Study
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Started | 12 | 7
Completed | 12 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (13.5) | 48.3 (12.9) | 40.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 8 | 2 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 7 | 19
Neurologic Level Number [Mean (Standard Deviation); unit: units on a scale] — The neurologic level number indicates the degree of neurologic functioning, with higher numbers indicating a higher degree of neurologic functioning. This is a continuous scale with 30 levels beginning at C1 (closest to the head) and moving caudal along the body to S5--C1 corresponds to level 1 and S5 corresponds to level 30.
  units on a scale | 7.7 (6.2) | 8.1 (5.3) | 7.8 (5.9)
Number of Days from Injury [Mean (Standard Deviation); unit: days] | 20.8 (9.3) | 19.9 (6.2) | 20.5 (8.3)
Admission Functional Independence Measure (FIM) motor subscale [Mean (Standard Deviation); unit: units on a scale] — The FIM motor subscale consists of 13 items: Eating, Grooming, Bathing, Dressing (upper body), Dressing (lower body), Toileting, Bladder management, Bowel management, Transfers (bed/chair/wheelchair), Transfers (toilet), Transfers (bath/shower), Walk/wheelchair, and Stairs. Each individual item is scored from 1 to 7. The range of total scores is 13 to 91, with a higher score indicating more independence in performing the task associated with each item.
  units on a scale | 16.7 (5.1) | 16.4 (5.6) | 16.6 (5.3)
Admission Functional Independence Measure (FIM) bladder item [Mean (Standard Deviation); unit: units on a scale] — The FIM bladder item (which is part of the FIM motor subscale) is scored from 1 to 7, with a range of possible scores from 1 to 7. A higher score indicates more independence in bladder management.
  units on a scale | 1 (0) | 1 (0) | 1 (0)
Admission Functional Independence Measure (FIM) cognition subscale [Mean (Standard Deviation); unit: units on a scale] — The FIM cognitive subscale consists of 5 items: Comprehension, Expression, Social interaction, Problem solving, and Memory. Each individual item is scored from 1 to 7. The range of total scores is 5 to 35, with a higher score indicating more independence in performing the task associated with each item.
  units on a scale | 27.8 (5.6) | 29.1 (5) | 28.3 (5.4)
Number of Participants with Tetraplegia [Count of Participants; unit: Participants] | 6 | 4 | 10
Number of Participants with American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade A [Count of Participants; unit: Participants] — Injuries are classified in as being neurologically "complete" or "incomplete" based "Sacral Sparing," which refers to the presence of sensory or motor function in the most caudal sacral segments as determined by the examination (i.e. preservation of light touch or pin prick sensation at the S4-5 dermatome, DAP or voluntary anal sphincter contraction). A complete injury is defined as the absence of sacral sparing, whereas an incomplete injury is defined as the presence of sacral.
  Grade A = Complete. No sensory or motor function is preserved in the sacral segments S4-S5.
  Participants | 8 | 3 | 11
American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade B [Count of Participants; unit: Participants] — See ASIA Grade A baseline measure description for further description of ASIA grading.
  Grade B = Sensory incomplete. Sensory but not motor function is preserved below the neurological level and includes the sacral segments S4-S5, AND no motor function is preserved more than three levels below the motor level on either side of the body.
  Participants | 2 | 1 | 3
American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade C [Count of Participants; unit: Participants] — See ASIA Grade A baseline measure description for further description of ASIA grading.
  Grade C = Motor incomplete. Motor function is preserved below the neurological level of injury, and more than half of key muscle functions below the single neurological level of injury have a muscle grade less than 3 (Grades 0-2).
  Participants | 2 | 2 | 4
American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade D [Count of Participants; unit: Participants] — See ASIA Grade A baseline measure description for further description of ASIA grading.
  D = Motor incomplete. Motor function is preserved below the neurological level of injury, and at least half (half or more) of key muscle functions below the neurological level of injury have a muscle grade >3.
  Participants | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infection
Description: All infections were urinary tract infections (UTIs).
Time Frame: about 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 12 | 7
Participants | 4 | 3

2. Primary Outcome: Number of Participants With Skin Irritation
Description: Number of participants with skin irritation, which includes cellulitis, burn, or pressure injury. The one instance of skin irritation was pressure injury.
Time Frame: about 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 12 | 7
Participants | 0 | 1

3. Primary Outcome: Number of Participants Who Were Unexpectedly Discharged to an Acute Care Hospital
Time Frame: about 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 12 | 7
Participants | 0 | 0

4. Primary Outcome: Mean Change in Pain Score as Indicated by Numeric Pain Scale (NPS)
Description: Participants received 30 minutes of TTNS (or sham stimulation) on each of 10 days over a 16-day period, and on each of the 10 days, pain was recorded immediately before stimulation (baseline) and at about 30 minutes later at the end of stimulation. For a single subject's "mean change in pain score": [Average of the post-stimulation measurements for all 10 time points] minus [Average of baseline measurements for all 10 time points time point] = [mean change in pain score]. The value reported is the mean of all participants' "mean change in pain score." The range of possible pain scores on the numeric pain scale is 1 to 10, with higher scores indicating higher level of pain.
Time Frame: baseline, about 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 12 | 7
units on a scale | -0.01 (0.22) | -0.06 (0.13)

5. Secondary Outcome: Maximum Detrusor Pressure as Evaluated by Urodynamic Study
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 12 | 7
cm H2O | 30.6 (21) | 33 (11.1)

6. Secondary Outcome: Maximum Detrusor Pressure as Evaluated by Urodynamic Study
Time Frame: 2 weeks
Population: One subject declined to repeat the post-TTNS urodynamic study, leaving 11 remaining in the TTNS group for the urodynamic measurements.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 11 | 7
cm H2O | 38.1 (21.4) | 44.4 (21.5)

7. Secondary Outcome: Maximum Bladder Capacity as Evaluated by Urodynamic Study
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 12 | 7
mL | 580 (45.7) | 571 (81.3)

8. Secondary Outcome: Maximum Bladder Capacity as Evaluated by Urodynamic Study
Time Frame: 2 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
Number analyzed (Participants) | 11 | 7
mL | 552.6 (110) | 459.6 (156.4)

ADVERSE EVENTS:
Time Frame: About 4 weeks
Arm/Group | Transcutaneous Tibial Nerve Stimulation | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7
Other Adverse Events (participants affected / at risk) | 4/12 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcutaneous Tibial Nerve Stimulation (N=12) | Control (N=7)
Deep Vein Thrombosis/Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 3 (3)
Pressure Injury (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT02573402/Prot_SAP_000.pdf